CLINICAL TRIAL: NCT00096148
Title: Randomized Phase II Trial of Idarubicin + Ara-C +/- Bevacizumab in Patients Age < 60 With Untreated Acute Myeloid Leukemia
Brief Title: Idarubicin and Cytarabine With or Without Bevacizumab in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02627; MDA-2004-0342; N01CM62202 (NIH); N01CM62204 (NIH); CDR0000391189 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Childhood Acute Basophilic Leukemia; Childhood Acute Eosinophilic Leukemia; Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Idarubicin; Cytarabine; Bevacizumab

ARMS (2):
- Arm I (idarubicin, cytarabine) (Experimental): Arm I: Patients receive idarubicin IV over 1 hour on days 1-3 and cytarabine IV continuously over 24 hours on days 1-4.
  Post-CR therapy: All patients receive 4 post-CR chemotherapy courses approximately every 28 days in the absence of disease progression or unacceptable toxicity.
  Course 1: Patients receive cytarabine IV continuously over 24 hours on days 1-5.
  Course 2 and 4: Patients receive idarubicin IV over 1 hour and cytarabine IV continuously over 24 hours on days 1-4.
  Interventions: Drug: idarubicin; Drug: cytarabine; Other: laboratory biomarker analysis
- Arm II (idarubicin, cytarabine, bevacizumab) (Experimental): Patients receive idarubicin and cytarabine as in arm I. Patients also receive bevacizumab* IV over 30-90 minutes on day 1. Patients who do not achieve complete remission (CR) after the first induction course may receive a second induction course approximately 28 days* later. Patients who do not achieve CR after 2 courses are removed from the study.
  NOTE: *Patients in arm II receive bevacizumab, independently of chemotherapy administration schedule, once every 21 days for 1 year from CR date.
  Post-CR therapy: All patients receive 4 post-CR chemotherapy courses approximately every 28 days in the absence of disease progression or unacceptable toxicity.
  Course 1: Patients receive cytarabine IV continuously over 24 hours on days 1-5.
  Course 2 and 4: Patients receive idarubicin IV over 1 hour and cytarabine IV continuously over 24 hours on days 1-4.
  Interventions: Drug: idarubicin; Drug: cytarabine; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm II (idarubicin, cytarabine, bevacizumab)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Bevacizumab may stop the growth of cancer by stopping blood flow to the leukemic cells in the bone marrow. Giving idarubicin and cytarabine with bevacizumab may kill more cancer cells. It is not yet know whether giving idarubicin together with cytarabine is more effective with or without bevacizumab in treating acute myeloid leukemia. This randomized phase II trial is studying how well giving idarubicin and cytarabine together with bevacizumab works compared to idarubicin and cytarabine alone in treating patients with newly diagnosed acute myeloid leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the activity of idarubicin and cytarabine with or without bevacizumab in patients with newly diagnosed acute myeloid leukemia.

II. Compare the proportion of patients who survive and remain in first complete remission (CR) one year from achieving CR after treatment with these regimens.

SECONDARY OBJECTIVES:

I. Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (< 45 vs 45 to 59), cytogenetics (normal vs -5/-7 vs other), flt 3 status (normal vs mutated), and type of acute myeloid leukemia (AML) (de novo vs secondary [arising after cytotoxic therapy or after an antecedent hematologic disorder, defined as a documented abnormality in blood count for >= 3 months before diagnosis of AML]. Patients who require treatment before cytogenetics or flt 3 status is known (e.g., patients with WBC > 50,000 OR with organ dysfunction thought to be due to blast infiltration) are stratified only according to age and type of AML. Induction therapy: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive idarubicin IV over 1 hour on days 1-3 and cytarabine IV continuously over 24 hours on days 1-4.

Arm II: Patients receive idarubicin and cytarabine as in arm I. Patients also receive bevacizumab* IV over 30-90 minutes on day 1. Patients who do not achieve complete remission (CR) after the first induction course may receive a second induction course approximately 28 days* later. Patients who do not achieve CR after 2 courses are removed from the study.

NOTE: *Patients in arm II receive bevacizumab, independently of chemotherapy administration schedule, once every 21 days for 1 year from CR date.

Post-CR therapy: All patients receive 4 post-CR chemotherapy courses approximately every 28 days in the absence of disease progression or unacceptable toxicity.

Course 1: Patients receive cytarabine IV continuously over 24 hours on days 1-5.

Course 2 and 4: Patients receive idarubicin IV over 1 hour and cytarabine IV continuously over 24 hours on days 1-4.

Course 3: Patients receive idarubicin IV over 1 hour and cytarabine IV continuously over 24 hours on days 1-2. After completion of the 4 post-CR chemotherapy courses, patients in arm I induction therapy do not receive further therapy. Patients in arm II induction therapy continue to receive bevacizumab as described above.After completion of study treatment, patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 60-120 patients (30-60 per treatment arm) will be accrued for this study within 12-30 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute myeloid leukemia (AML)

  * No acute promyelocytic leukemia
  * None of the following cytogenetic abnormalities*:

    * t(8;21)
    * t(16;16)
    * inv(16)
* No history or clinical evidence of primary brain tumors or brain metastasis
* Performance status - ECOG 0-2
* No bleeding diathesis or coagulopathy (unless related to AML)
* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 times ULN
* No proteinuria
* No more than 1 g of protein on 24-hour urine collection
* LVEF ≥ 50%
* No uncontrolled hypertension
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No peripheral vascular disease ≥ grade II
* No stroke within the past 6 months
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Myocardial infarction
  * Unstable angina
* No other clinically significant cardiovascular disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3-4 months after study participation
* No serious or non-healing wound ulcer or bone fracture
* No uncontrolled infection
* No significant traumatic injury within the past 28 days
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history or clinical evidence of CNS disease (e.g., seizures not controlled with standard medical therapy)
* Prior or concurrent transfusions or hematopoietic growth factors for AML allowed

  * No concurrent prophylactic hematopoietic colony-stimulating factors
* Prior or concurrent hydroxyurea for AML allowed
* More than 28 days since prior major surgery or open biopsy
* No concurrent major surgery
* No other prior therapy for AML
* No concurrent full-dose anticoagulation therapy

  * Concurrent prophylactic anticoagulation (e.g. low-dose warfarin to maintain patency of permanent indwelling IV catheters) allowed provided INR < 1.5
* No other concurrent anticancer therapies
* No other concurrent investigational cytotoxic agents

Max Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2004-10; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who remain alive in the first complete remission (CR) 1 year from achievement of CR assessed every 3 weeks for 1 year | 13 months from registration
  Fisher's exact test will be used to compare the proportion of patients alive in CR 13 months from registration date. The test has approximately 89% power to detect an absolute increase of 20% in this proportion, testing at the one-sided 0.15 significance level.

SECONDARY OUTCOMES:
Safety of idarubicin+cytarabine+bevacizumab by AdEERS, CBC and chem. | Up to 2 years after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States